CLINICAL TRIAL: NCT03782402
Title: The Effect of Dispensed Cannabis on Taxane Induced Peripheral Neuropathy
Brief Title: Cannabinoids for Taxane Induced Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding being sought
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Psychiatrist II, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7635
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Cannabinoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabinoids (THC and CBD) (Experimental): THC and CBD
  Interventions: Drug: Cannabinoids
- Placebo Cannabinoids (Placebo Comparator): placebo cannabinoids
  Interventions: Drug: Cannabinoids

INTERVENTIONS:
Drug: Cannabinoids — Cannabinoids with THC and CBD versus placebo cannabinoids

SUMMARY:
Taxane-induced peripheral neuropathy (TIPN) affects a significant number of women undergoing breast cancer treatment. Some patients may need to shorten their course of treatment, and do not receive the full benefit of chemotherapy as a result. Rodent studies have shown that the cannabinoids may significantly improve hyperalgesia and allodynia induced by paclitaxel. The goal of this study is to investigate the cannabinoids THC and CBD for TIPN.

DETAILED DESCRIPTION:
The investigators' goal is to study the efficacy of cannabinoids as a potential treatment for TIPN. Volunteers with a diagnosis of breast cancer and chemotherapy-induced peripheral neuropathy, secondary to treatment with paclitaxel or docetaxel, will be enrolled. This study involves the administration of cannabinoids in different strength capsules. The primary outcome measures include measures of pain and functional impairment (non-painful symptoms). The scales will include: 1) Brief Pain Inventory-Short Form (BPI) for pain severity ; and 2) BPI pain interference subscale for functional impairment. The study outcomes will also include secondary measures of perception, which will be performed in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* 1) Participants with breast cancer, experiencing TIPN due to paclitaxel or docetaxel.
* 2) Participants must have an ECOG score of 2 or better. Participants must have a score of 2 or 3 score for sensory neuropathy, as assessed by the Common Toxicity Criteria Adverse Events (CTCAE).
* 3) Able to give informed consent and comply with all study procedures.

Exclusion Criteria:

* 1) Diagnosis of a major medical, neurological, or psychiatric disorder that would preclude study participation.
* 2) Women who are not practicing an effective form of birth control (condoms, diaphragm, birth control pill, IUD) or currently pregnant.
* 3) Subjects taking warfarin.
* 4) Subjects with orthostatic hypotension, hypertension, cardiovascular disease, or neurodegenerative disorders.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned based on history of cannabis use.
Groups:
- Cannabinoids (THC and CBD): Cannabinoids with THC and CBD, titrated to a maximum of 15 mg THC, 300 mg CBD
- Placebo Cannabinoids: Placebo cannabinoids for comparison
Period: Overall Study
Arm/Group | Cannabinoids (THC and CBD) | Placebo Cannabinoids
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cannabinoids (THC and CBD): Cannabinoids THC and CBD titrated
- Total: Total of all reporting groups
Arm/Group | Cannabinoids (THC and CBD) | Placebo Cannabinoids | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8) | 54 (8) | 54 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 3 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory-Short Form (BPI)
Description: This is a standard questionnaire to measure pain.It is used to evaluate pain through a number of different scales. Patients fill out 11 different questions that ask about pain intensity (present and least, most, and average for the past 24 hours) and the effect of the pain on the ability to function during various activities of daily living. Higher number is worse. range is 0 to 10
Time Frame: value at the later time (8 weeks) point minus the value at the earlier time point (baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cannabinoids (THC Ans CBD): Cannabinoids with different concentrations of THC and CBD
- Placebo Cannabinoids: Placebo with no THC to CBD
Arm/Group | Cannabinoids (THC Ans CBD) | Placebo Cannabinoids
Number analyzed (Participants) | 6 | 6
units on a scale | 4.8 (1.5) | 5.8 (1.5)

2. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy Taxane
Time Frame: Baseline and weekly until end of study.
Reporting Status: Not Posted, anticipated posting 2028-10

3. Post Hoc Outcome: Total Neuropathy Score (TNSc) a Scale of Sensory, Motor and Autonomic Symptom
Time Frame: Baseline and weekly until end of study
Reporting Status: Not Posted, anticipated posting 2030-10

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 8 weeks.
Description: No participants were expected to ne at risk for all-cause mortality.
Groups:
- Cannabinoids (THC and CBD); Placebo Cannabinoids: Strengths of cannabinoids will vary across groups
  Cannabinoids: Cannabinoids with different concentrations of THC and CBD
Arm/Group | Cannabinoids (THC and CBD) | Placebo Cannabinoids
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabinoids (THC and CBD) (N=6) | Placebo Cannabinoids (N=6)
Sedation (Nervous system disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Please note: this was a pilot study that was not funded for a full study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT03782402/Prot_SAP_ICF_000.pdf